CLINICAL TRIAL: NCT02779556
Title: Health Literacy Intervention to Improve Diabetes Outcomes Among Rural Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Northwestern University (Other); Louisiana State University Health Sciences Center Shreveport (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204290; 1R01DK107572-01A1 (NIH)
Record Dates: First submitted 2016-05-04; First posted 2016-05-20 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Diabetes
Keywords: Health Literacy; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Other): ADA Living Well with Diabetes Workbook, 15 minute in-person counseling, follow-up every 3 months
  Interventions: Other: ADA Living Well with Diabetes Workbook
- Intervention (Other): ACP Living with Diabetes Guide, 15 minute in-person counseling , 15 minute follow-up counseling (3, 6, and 9 months), monthly phone calls after 3 months
  Interventions: Other: ACP Living with Diabetes Guide

INTERVENTIONS:
Other: ACP Living with Diabetes Guide — American Colleges of Physicians (ACP) Living Well with Diabetes Guide
  Arms: Intervention
Other: ADA Living Well with Diabetes Workbook — American Diabetes Association (ADA) Living Well with Diabetes Workbook
  Arms: Enhanced Usual Care

SUMMARY:
The researchers will conduct a patient-randomized, pragmatic clinical trial among 6 rural PCMHs in Arkansas, targeting individuals with uncontrolled type 2 diabetes.

The primary aims are to:

1. test the effectiveness of the ACP diabetes health literacy intervention to improve a range of diabetes-related outcomes among rural patients;
2. compared to usual care, evaluate whether the intervention reduces disparities by patient literacy level.

   The secondary aims are to:
3. investigate whether a threshold or gradient effect exists between the amount of follow-up counseling (number of action plans) and intervention effectiveness;
4. determine the fidelity of all intervention components, and explore any identified patient, provider (physician, nurse, health coach), and/or health system barriers to implementation; and
5. assess the costs associated with implementing the intervention from a health system perspective.

DETAILED DESCRIPTION:
The investigators will test the effectiveness and fidelity of embedding the American College of Physicians (ACP) diabetes health literacy intervention among patient-centered medical homes throughout rural Arkansas. Proper diabetes self-care requires patients to have considerable knowledge, a range of skills, and to sustain multiple health behaviors. Self-management interventions are needed that have been designed for individuals with lower literacy skills, that can be readily implemented and sustained among rural clinics with limited resources that disproportionately care for patients with limited literacy. Researchers on the team developed an evidence-based, patient-centered, low literacy ACP intervention promoting diabetes self-care that includes:

1. a diabetes guide that uses plain language and descriptive photographs to teach core diabetes concepts and empower patients to initiate behavior change;
2. a brief counseling strategy to assist patients in developing short-term, explicit and attainable goals for behavior change ('action plans');
3. a training module for physicians, nurses, and medical assistants that prepares providers to assume educator/counselor roles with the Diabetes Guide as a teaching tool;
4. electronic tracking and monitoring tools for primary care practices.

While the intervention has previously been field tested and found to significantly improve patient knowledge, self-efficacy, and engagement in related health behaviors, it has not yet been comprehensively tested in practices, and its optimal implementation is not known. The investigators now have a unique opportunity to learn from prior evaluation, modify and disseminate an ACP health literacy intervention among patients with type 2 diabetes cared at rural clinics in Arkansas that are Patient-Centered Medical Homes (PCMH). These practices are embedding care coordination services that can be leveraged to improve chronic disease management. All are supervised by a new University of Arkansas for Medical Sciences (UAMS) Center for Health Literacy. The investigators' revised intervention will blend outsourced and clinic-based approaches and redeploy health coaches for counseling self-management mostly via phone, but also at the point-of-care. This is a feasible way to reach rural, vulnerable patients. The investigators will conduct a patient-randomized, pragmatic clinical trial among 6 rural PCMHs in Arkansas, targeting individuals with uncontrolled type 2 diabetes.

The primary aims are to:

1. test the effectiveness of the ACP diabetes health literacy intervention to improve a range of diabetes-related outcomes among rural patients;
2. compared to usual care, evaluate whether the intervention reduces disparities by patient literacy level.

   The secondary aims are to:
3. investigate whether a threshold or gradient effect exists between the amount of follow-up counseling (number of action plans) and intervention effectiveness;
4. determine the fidelity of all intervention components, and explore any identified patient, provider (physician, nurse, health coach), and/or health system barriers to implementation; and
5. assess the costs associated with implementing the intervention from a health system perspective.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* English speaking
* active patient at regional family medical center study site
* confirmed diagnosis of type 2 diabetes as documented in the electronic health record
* recent Hemoglobin A1c reading of >7.5% and less than or equal to 10%

Exclusion Criteria:

* uncorrectable visual impairments
* hearing impairments
* cognitive impairments

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Hadden, PhD, Principal Investigator — University of Arkansas
Locations (6):
- United States (6):
  - UAMS Family Medical Center Northwest, Fayetteville, Arkansas
  - UAMS Family Medical Center Fort Smith, Fort Smith, Arkansas
  - UAMS Family Medical Center Jonesboro, Jonesboro, Arkansas
  - UAMS Family Medical Center Magnolia, Magnolia, Arkansas
  - UAMS Family Medical Center Pine Bluff, Pine Bluff, Arkansas
  - UAMS Family Medical Center Texarkana, Texarkana, Arkansas

IPD SHARING:
Plan to Share IPD: Yes
The investigators are committed to the open and timely dissemination of the research outcomes. Plans for sharing resources with the scientific community include presentations and publications in peer-reviewed journals. The final data set will be made available to NIH investigators upon request. Consulting with program officer to ensure data sharing compliance.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This will be available 6 months after publication of main study results.
Access Criteria: Require an NIH investigator with an IRB approved protocol, to conduct secondary data analysis of the available dataset.

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Enhanced Usual Care | Intervention
Started | 394 | 362
Completed | 393 | 362
Not Completed | 1 | 0
Not completed — Partial baseline interview completed | 1 | 0
Period: 3 Months
Arm/Group | Enhanced Usual Care | Intervention
Started | 393 | 362
Completed | 326 | 314
Not Completed | 67 | 48
Not completed — Lost to Follow-up | 40 | 29
Not completed — Missed 3 month clinic visit | 27 | 19
Period: 6 Month
Arm/Group | Enhanced Usual Care | Intervention
Started | 353 (Those who were not lost to follow-up but missed the visit from the previous period were allowed to continue in the study and complete future interviews (314+19=333 Enhanced Usual Care).) | 333 (Those who were not lost to follow-up but missed the visit from the previous period were allowed to continue in the study and complete future interviews (326+27=353 Intervention).)
Completed | 320 | 294
Not Completed | 33 | 39
Not completed — Lost to Follow-up | 33 | 39
Period: 6 Month HbA1c
Arm/Group | Enhanced Usual Care | Intervention
Started | 394 (All enrolled participants were eligible for the analysis of clinical values regardless of completion of 3 and 6 month interviews.) | 362 (All enrolled participants were eligible for the analysis of clinical values regardless of completion of 3 and 6 month interviews.)
Completed | 325 | 312
Not Completed | 69 | 50
Not completed — No value collected during window | 69 | 50
Period: 12 Month HbA1c
Arm/Group | Enhanced Usual Care | Intervention
Started | 394 (All enrolled participants were eligible for the analysis of clinical values regardless of completion of 3 and 6 month interviews.) | 362 (All enrolled participants were eligible for the analysis of clinical values regardless of completion of 3 and 6 month interviews.)
Completed | 256 | 260
Not Completed | 138 | 102
Not completed — No value collected during window | 138 | 102

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | Intervention | Total
Number analyzed (Participants) | 394 | 362 | 756
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (11.8) | 56.1 (11.4) | 55.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 235 | 510
  Male | 119 | 127 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 388 | 353 | 741
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 220 | 191 | 411
  White | 166 | 160 | 326
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 1 | 3 | 4
Education [Count of Participants; unit: Participants]
  Less than High School | 87 | 66 | 153
  High School Graduate | 141 | 127 | 268
  Some College | 126 | 117 | 243
  College Graduate | 40 | 50 | 90
  Refused to answer question | 0 | 2 | 2
Health Literacy (NVS) [Count of Participants; unit: Participants] — Health Literacy (NVS) Newest Vital Sign
  Participants
    Limited | 210 | 183 | 393
    Adequate | 184 | 179 | 363

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C (HbA1C)
Description: HbA1C will be obtained from patients' electronic health records, defined as the value closest to 6 months post baseline. The hemoglobin A1c (HbA1c) value ranges from approximately 4 to 14% where higher HbA1c value means worse outcome.
Time Frame: Six months
Population: 119 individuals were excluded from analysis, because they did not have a 6 month HbA1c value within the designated window.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of glycated hemoglobin
Arm/Group | Enhanced Usual Care | Intervention
Number analyzed (Participants) | 325 | 312
Percentage of glycated hemoglobin | 8.4 [8.3 to 8.6] | 8.3 [8.1 to 8.5]

2. Primary Outcome: Hemoglobin A1C (HbA1C)
Description: HbA1C will be obtained from patients' electronic health records, defined as the value closest to 12 months post baseline. The hemoglobin A1c (HbA1c) value ranges from approximately 4 to 14% where higher HbA1c value means worse outcome.
Time Frame: Twelve months
Population: 240 individuals were excluded from analysis, because they did not have a 12 month HbA1c value within the designated window.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of glycated hemoglobin
Arm/Group | Enhanced Usual Care | Intervention
Number analyzed (Participants) | 260 | 256
Percentage of glycated hemoglobin | 8.5 [8.3 to 8.7] | 8.4 [8.2 to 8.6]

3. Secondary Outcome: Diabetes Knowledge
Description: A self-reported Diabetes Knowledge Questionnaire that uses 13 multiple choice questions will be administered. Total scores range from 0-13 where higher scores demonstrate more knowledge.
Time Frame: Three months
Population: 116 participants were excluded, missed 3 month visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Enhanced Usual Care | Intervention
Number analyzed (Participants) | 326 | 314
Score on a scale | 9.2 [9.0 to 9.4] | 9.3 [9.1 to 9.5]

4. Secondary Outcome: Diabetes Knowledge (0-13)
Description: as for outcome 3
Time Frame: Six months
Population: 142 participants were excluded, missed 6 month visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Enhanced Usual Care | Intervention
Number analyzed (Participants) | 320 | 294
Score on a scale | 9.5 [9.3 to 9.6] | 9.7 [9.5 to 9.9]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Enhanced Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 6/394 | 3/362
Serious Adverse Events (participants affected / at risk) | 0/394 | 0/362
Other Adverse Events (participants affected / at risk) | 0/394 | 0/362

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT02779556/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT02779556/ICF_001.pdf